CLINICAL TRIAL: NCT03261453
Title: A Randomized, Multi-Center, Phased, Pivotal Safety and Efficacy Study Comparing the Elipse™ Gastric Balloon System vs. Sham for the Treatment of Obese Adults
Brief Title: THE ENLIGHTEN STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allurion Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRL-1000-0002
Record Dates: First submitted 2017-05-03; First posted 2017-08-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): Patients randomized to treatment will receive the Elipse device.
  Interventions: Device: Active Elipse Device
- Control (Sham Comparator): Patients randomized to the control arm will receive the sham device.
  Interventions: Device: Elipse Sham Device

INTERVENTIONS:
Device: Active Elipse Device — Intervention Device
  Other Names: Elipse Gastric Balloon System (active)
  Arms: Treatment
Device: Elipse Sham Device — Control Device
  Other Names: Elipse Gastric Balloon System (control)
  Arms: Control

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of the Elipse Gastric Balloon System for the treatment of obese adults.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, randomized, two-phase study to be conducted in a planned 400 obese individuals drawn from up to 15 sites. The treatment duration of the study is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years and ≤ 65 years of age
2. BMI ≥30 kg/m2 and ≤ 40 kg/m2
3. Have signed study specific Informed Consent Form
4. Willing to comply with study requirements, including follow-up visits
5. Documented negative pregnancy test in women of childbearing potential.
6. Women of childbearing potential not intending to become pregnant for the duration of study participation. (Note: Women of childbearing potential must not be nursing at the time of treatment).
7. Fully ambulatory without any severe chronic orthopedic disease that requires reliance on crutches, walkers or a wheelchair that could preclude exercise during the study.
8. Confirmed unsuccessful attempts at more conservative weight reduction alternatives, such as supervised diet, exercise and behavior modification programs attempted within the 24 months preceding enrollment.

Exclusion Criteria:

1. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease
2. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer
3. Previous bariatric or gastric surgery or likely to undergo during study
4. Use of an intragastric device prior to this study
5. Chronic pancreatitis or acute pancreatitis within 12 months of enrollment
6. History of or current small bowel obstructions
7. History of abdominal and/or pelvic surgery EXCLUDING only ONE of the following surgeries that was performed at least 12 months prior to study enrollment: cesarean section, diagnostic laparoscopy, laparoscopic appendectomy, laparoscopic cholecystectomy. (For example: if a patient has had 2 cesarean sections, or one cesarean section and a laparoscopic appendectomy, she would be excluded. If a patient had one cesarean section, she may be included)
8. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma) or immunocompromised
9. History of genetic or endocrine causes of obesity not adequately controlled by medication
10. History of/or signs and/or symptoms of/or radiographic evidence of esophageal, gastric, or duodenal disease including but not limited to hiatal hernias greater than or equal to 2 centimeter (cm), paraesophageal hernias, inflammatory diseases, cancer, varices, diverticula, gastroparesis, ulcers, stricture/stenosis, achalasia and esophagitis
11. Insulin-dependent diabetes (either Type 1 or Type 2)
12. Significant acute and/or chronic infections of any kind
13. Severe coagulopathy, hepatic insufficiency or cirrhosis
14. Unable or unwilling to discontinue use of aspirin and/or non-steroidal anti-inflammatory agents (NSAIDs) at least 14 days prior to Elipse Deployment and continuing for 14 days after Elipse excretion
15. Currently taking the following medications (within 30 days prior to enrollment) and/or there is a need or anticipated need for these medications during the study:

    Excluded Medications:

    Systemic corticosteroids Anticoagulant therapy (e.g. warafin, dabigatran) or anti-platelet therapy) Immunosuppressive therapy (e.g. azathioprine, cyclosporine) Prescription or over the counter weight loss medication(s) Medications known to cause significant weight gain or weight loss Narcotics, opiates or benzodiazepines Insulin for treatment of diabetes Anti-seizure therapy (e.g. clonazepam, phenytoin) Anti-arrhythmics (e.g. amidarone)
16. History of pulmonary embolism
17. Has cardiac pacemaker or other electric implantable device
18. Anemia defined as either:

    1. Hgb < 11 for females, <12 for males
    2. Abnormal red cell indices and iron deficiency
19. Smoking cessation within 3 months of enrollment or plans to quit smoking during the study
20. Documented total body weight loss of ≥ 5% anytime 6 months preceding enrollment
21. Residing in a location without ready access to study site medical resources
22. Inability to walk 200 yards without assistance
23. Eating disorders including night eating syndrome (NES), bulimia, or binge eating disorder
24. Unwilling to refrain from any reconstructive and/or cosmetic surgery that may affect body weight during the study such as mammoplasty and lipoplasty
25. Current or history of illicit drug use or excessive alcohol use
26. Enrolled in another investigational study that has not completed the required primary endpoint follow-up period (Note: Subjects involved in a long-term surveillance phase of another study are eligible for enrollment in this study).
27. Any conditions that, in the opinion of the investigator, may render the subject unable to complete the study with a likely fatal outcome, or lead to difficulties for subject compliance with study requirements, or could confound study data.
28. Patient is not of sufficient medical health as determined by the Investigator to participate in the study.
29. Employees/family members of Allurion Technologies or any of its affiliates or contractors
30. Immediate employees/family members of the Investigator, sub-Investigators, or their medical office or practice, or surgical, bariatric or hospital organizations at which study procedures may be performed
31. An immediate family member (by marriage or blood relationship) of another subject already enrolled in the study
32. Positive breath test for H. Pylori
33. History of or current inflammatory bowel disease (e.g. Crohn's disease, Ulcerative Colitis)

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Co-Primary Effectiveness Endpoint: Total Body Weight Loss (TBWL) Comparison Between Treatment and Control Group at 16 weeks | 16 weeks
  An inferential test of whether the Treatment Group Responder Rate (RR) dichotomized at 5% TBWL at 16 weeks is significantly greater than 35%.
Co-Primary Effectiveness Endpoint 2: Percent of Total Body Weight Loss (TBWL) Comparison Between Treatment and Control group | 16 weeks
  An inferential test of whether the Treatment Group mean %TBWL is significantly greater than Control Group mean % TBWL at 16 weeks
Primary Safety Endpoint: Incidence of overall procedure or device related Serious Adverse Events | 24 weeks
  The primary safety endpoint of this clinical investigation is the overall incidence of procedure- or device-related Serious Adverse Events through 24 weeks.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Honor Health, Scottsdale, Arizona
  - University of Colorado, Anschutz Health and Wellness Center, Aurora, Colorado
  - Bariatric Institute of Greater Chicago, Bolingbrook, Illinois
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - Holyoke Medical Center, Holyoke, Massachusetts
  - Weill Cornell Medicine, Division of Endocrinology, Diabetes and Metabolism, New York, New York
  - University of Pennsylvania Medical Center (UPMC), Pittsburgh, Pennsylvania
  - CHI Metabolic and Bariatric Care, Chattanooga, Tennessee
  - MidSouth Bariatrics, Memphis, Tennessee
  - Vanderbilt Center for Surgical Weight Loss, Nashville, Tennessee
  - UT Physicians Minimally Invasive Surgeons of Texas (UTMIST), Bellaire, Texas
  - Charlottesville Medical Research Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided